CLINICAL TRIAL: NCT06633263
Title: Combined Effect of Cognitive Behavioral Therapy for Insomnia and a Behavioral Activation Program for Depression on Depressive Symptoms and Insomnia : A Multiple Case Study
Brief Title: Combined Effect of TCC-I and BATD on Depressive Symptoms and Insomnia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Audrey Krings, Principal Investigator, University of Liege
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-313
Record Dates: First submitted 2024-10-02; First posted 2024-10-09 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Depression - Major Depressive Disorder; Insomnia
Keywords: depression; insomnia; CBT-I; BATD; combined intervention; multiple case study; Single Case Experimental Design
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: In condition 1 : CBT-I precede BATD In condition 2 : BATD precede CBT-I Condition 1 is starting in Novembre Condition 2 is starting in February
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I followed by BATD (Experimental): 1. Five group CBT-I sessions of two hours, one per week.
  2. Two-week break - baseline
  3. Five individual BATD sessions of one hour, one per week. Because of the diverse content of ruminations and avoidances in depression (Blairy et al., 2020), AC therapy will be administered in an individual format, while CBT-I will take place in a group setting.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Behavioral Activation Treatment for Depression
- BATD followed by CBT-I (Experimental): 1. Five individual BATD sessions of one hour, one per week. Because of the diverse content of ruminations and avoidances in depression (Blairy et al., 2020), AC therapy will be administered in an individual format, while CBT-I will take place in a group setting.
  2. Two-week break - baseline
  3. Five group CBT-I sessions of two hours, one per week.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Behavioral Activation Treatment for Depression

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Introduce self-recording with the sleep diary; Introduce basic notions of insomnia; Introduce basic notions of sleep hygiene; Introduce basic notions of sleep; Recreate a time and place dedicated to sleep; Limit time spent in bed to time slept; Promote attitudes and beliefs that favor sleep and manage worries; Relapse prevention. This intervention is empirically validated (Morin, 2022).
Behavioral: Behavioral Activation Treatment for Depression — Introduce self-recording with daily activities; Introduce the basic concept of depression; Identify and increase activities associated with positive reinforcement; Reflect on life domains and values to identify reinforcing activities; Identify and decrease activities associated with negative reinforcement; Identify and decrease activities associated with negative reinforcement; Relapse prevention. This intervention is empirically validated (Ciharova et al., 2021)

SUMMARY:
The goals of this interventional study is to study if the combine effects of Behavioral Activation Treatment for Depression (BATD) and Cognitive Behavioral Therapy for Insomnia (CBT-I) is effective on primary outcomes : depression, insomnia, well-being and anxiety and secondary outcomes : worry, rumination, behavioral inertia, experiential avoidance, anticipatory pleasure deficits, cognitive resource deficits, emotional reactivity, quality of sleep, and sleep beliefs for participants suffering from depression and insomnia disorders.

DETAILED DESCRIPTION:
Depression is a widespread mental disorder characterized by affective, cognitive and physiological disturbances that impact individuals' daily functioning. Sleep difficulties are an essential component of the clinical picture of depression. Several interventional studies have demonstrated the value of specific insomnia treatment in the management of depression. Indeed, the absence of targeted treatment for insomnia increases the risk of depressive relapse. In this context, the importance of specific treatment of insomnia in cases of comorbidity with depression, and the need to integrate this approach into clinical practice, have recently been highlighted. However, very few studies have explored the efficacy of combined treatment of insomnia (with Cognitive Behavioural Therapy for Insomnia - CBT-I) and depression (with Behavioural Activation Treatment for Depression - BATD). However, one study has shown that BATD can have beneficial effects on sleep quality (in caregivers of people with Alzheimer's disease). The combined treatment of CBT-I and BATD, as well as the importance of the order of administration of these interventions in cases of insomnia-depression comorbidity, however, remain unexplored.

The aim of this study is to evaluate the overall effect of the combination of CBT-I and a BATD on depressive symptoms and insomnia in the short, medium and long term. It also seeks to examine the specific effects of each intervention. In addition, the study assesses efficacy and adherence under two different orders of treatment combination, while exploring the psychological mechanisms likely to promote positive symptoms change. Finally, it looks at inter-individual differences in responses to interventions. Our study will help provide empirical evidence on the efficacy of combined treatment for people suffering from insomnia and depression. By identifying the psychological mechanisms that may promote improvement in these comorbid disorders, it could also help refine and improve current treatments.

Participants will be recruited through a number of sources, including the CPLU (Clinique Psychologique et Logopédique de l Université de Liège), word of mouth, announcements within the University (e.g. via the student and staff quality of life service), social networks, and various CHU departments. A flyer will be distributed by clinicians and on social networks, including Facebook. Participants will also be identified through CHU psychologists, doctors and psychiatrists, who have potential access to the target population (people suffering from sleep disorders and depression).

An initial telephone interview will take place to check the inclusion and exclusion criteria, explain how the study works and the various appointment dates.

Participants wishing to take part in the study, but presenting exclusion criteria, will be redirected to appropriate care services according to their difficulties. This may include services specializing in sleep disorders, services dedicated to the management of psychological disorders, psychiatric emergencies in the event of significant suicidal ideation, or individual psychological follow-up by a specialized therapist (such as primary care psychologists or CBT psychotherapists).

If the person meets the criteria, an initial interview will be arranged. During this first clinical interview, the protocol will be presented in greater detail. Participants' expectations and motivations will be investigated to ensure that the proposed intervention can meet them. The information letter and informed consents will be offered to the participant. A socio-demographic questionnaire will be proposed. The content of the assessments to be completed daily will be presented to the participants. At the end of this interview, they will also be invited to complete the standardized pre-intervention questionnaires.

Participants will then begin self-observation for two weeks, before starting the first intervention (CBT-I in condition 1 and BATD in condition 2). This will be followed by a further two-week period of observation without intervention, prior to the second intervention (BATD in condition 1 and CBT-I in condition 2). A final two-week self-observation phase follows the second intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults with depression (PhQ 9 > 10; cut-off for moderate depression) and insomnia (Insomnia Severity Index > 11) who also meet DSM-V criteria for depression and insomnia (APA, 2013) and have a good understanding of French.

Exclusion Criteria:

* Participants requiring different treatment, i.e. those with symptoms suggestive of psychotic disorder, bipolar disorder, substance abuse disorder, excessive suicidal ideation, or other sleep pathology (such as sleep apnea, restless legs syndrome, narcolepsy, sleepwalking, or periodic limb movements)
* Participants who have recently received or are currently receiving other interventions that could be confused with our intervention, such as those undergoing treatment for sleep or depression, or those undergoing parallel psychological or pharmacological treatment (antidepressants and anxiolytics will be accepted provided they have been stabilized for at least two months and there are no planned changes in the following weeks).
* Participants with commitments that disrupt nocturnal sleep cycles and habits, such as those who no longer work or who work night shifts, will also be excluded from the study.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Six measures. Up to two weeks before the intervention, up to two weeks after the first intervention, up to two weeks after the second intervention, three months after the second intervention, six months after the second intervention, and two years after
  Generalised Anxiety Disorder Questionnaire. Scores ranges from 0 to 21. Higher scores means worse outcome (higher anxiety symptoms)
Depression | Six measures. Up to two weeks before the intervention, up to two weeks after the first intervention, up to two weeks after the second intervention, three months after the second intervention, six months after the second intervention, and two years after
  Patient Health Questionnaire. Scores ranges from 0 to 27. Higher scores means worse outcome (higher depressive symptoms)
Insomnia | Six measures. Up to two weeks before the intervention, up to two weeks after the first intervention, up to two weeks after the second intervention, three months after the second intervention, six months after the second intervention, and two years after
  Insomnia Severity Index. Scores ranges from 0 to 28. Higher scores means worse outcome (higher insomnia)
Fatigue | Six measures. Up to two weeks before the intervention, up to two weeks after the first intervention, up to two weeks after the second intervention, three months after the second intervention, six months after the second intervention, and two years after
  Multidimensional Fatigue Inventory - General and physical fatigue. Scores ranges from 9 to 45. Higher scores means worse outcome (higher general and physical fatigue).
Well-being | Six measures. Up to two weeks before the intervention, up to two weeks after the first intervention, up to two weeks after the second intervention, three months after the second intervention, six months after the second intervention, and two years after
  Well-being - Warwick-Edinburgh Mental Wellbeing Scale. Scores ranges from 14 to 70. Higher scores means better outcome (higher well-being)
Socio-démographic Questionnaires | Up to two weeks before the intervention
  Age, gender, socio-economical status, situation at home

SECONDARY OUTCOMES:
Sleep Beliefs | Six measures. Up to two weeks before the intervention, up to two weeks after the first intervention, up to two weeks after the second intervention, three months after the second intervention, six months after the second intervention, and two years after
  Dysfunctional Beliefs and Attitudes about Sleep Scale. Scores ranges from 0 to 160. Higher scores means worse outcome (higher dysfunctional beliefs)
Client satisfaction | Two measures. up to two weeks after the first intervention, up to two weeks after the second intervention,
  Consumer Satisfaction Questionnaire. Scores ranges from 8 to 32. Higher scores means better outcome (higher satisfaction)
Activation | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Activation level was collected daily at the end of the day in a booklet with the following item -I have been an active person and have accomplished the goals I set for myself- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means better outcome (higher behavioral activation)
Rumination | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Rumination level was collected daily at the end of the day in a booklet with the following item -I spent a lot of time dwelling on my problems- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means worse outcome (higher rumination)
Anticipatory pleasure | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Anticipatory pleasure level was collected daily at the end of the day in a booklet with the following item -I m looking forward to some upcoming events or activities- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means better outcome (higher anticipatory pleasure)
Avoidance | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Avoidance level was collected daily at the end of the day in a booklet with the following item -Most of the things I did were aimed at escaping or avoiding something unpleasant.- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means worse outcome (higher avoidance)
Worry | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Worry level was collected daily at the end of the day in a booklet with the following item -I worry about everything all the time- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means worse outcome (higher worry)
Emotional reactivity | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Emotional Reactivity level was collected daily at the end of the day in a booklet with the following item -I have found it difficult to cope emotionally with stressful situations or events that others might consider unimportant- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means worse outcome (higher emotional reactivity)
Emotional reactivity 2 | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Emotional Reactivity 2 level was collected daily at the end of the day in a booklet with the following item -I have a tendency to react strongly, emotionally, to stressful situations or events that could have a negative impact on my sleep- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means worse outcome (higher emotional reactivity)
Cognitive ressources - Focusing | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Cognitive ressources level was collected daily at the end of the day in a booklet with the following item -It was easy for me to concentrate on a difficult task, even when there was noise all around- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means better outcome (better attentional focusing).
Cognitive ressources - Flexibility | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Cognitive ressources level was collected daily at the end of the day in a booklet with the following item -It was easy for me to alternate between two different tasks- accompanied by a visual Analogue Scale (ranging from left side : not at all to right side completely). Scores ranges from 0 to 10. Higher scores means better outcome (better attentional flexibility)
Sleep quality | Everyday through intervention completion (from week 1 up to 16 weeks later)
  Sleep quality (Sleep onset latency, Total sleep Time, Wake after sleep onset, sleep efficiency) was collected daily via a sleep diary. Higher sleep onset latency and higher wake after sleep onset scores means a worse outcome, higher total sleep time and sleep efficiency means a better outcome

OTHER OUTCOMES:
Qualitative Interview | Three measures. Up to two weeks before the intervention, up to two weeks after the first intervention, up to two weeks after the second intervention
  A semi-structured interview with open-ended questions focusing on participants; experiences and change processes.

CONTACTS AND LOCATIONS:
Locations (1):
- CPLU (clinique psychologique et logopédique de l université de Liège), Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: CSR
Time Frame: Beginning after publication with no end date
Access Criteria: meta-analysis and that must be approved by the investigator

REFERENCES:
- See also: pré-registration and data — https://osf.io/dhmj8/
- Available data/document: Study Protocol — https://osf.io/dhmj8/
- Available data/document: Individual Participant Data Set — https://osf.io/dhmj8/